CLINICAL TRIAL: NCT07188948
Title: In Vivo Cross-Modal Imaging of Skin - VISION2
Brief Title: In Vivo Cross-Modal Imaging of Skin
Acronym: VISION2
Status: Recruiting | Type: Observational
Sponsor: Gabriel Sanchez (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gabriel Sanchez, CEO, Enspectra Health
Organization: Enspectra Health (Industry)
Other Study IDs: CR-30359; 5R44CA285138-02 (NIH)
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Skin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Skin conditions — Participants with skin conditions such as AK or participants without any skin conditions (healthy skin)
Device: Skin Condition — Participants with Skin conditions or participants without any skin conditions (Healthy)

SUMMARY:
The overall objective of this study is to use VIO/FG-30350 ("VIO") to observe microscopic skin structure in people of different skin health at different anatomic locations and correlate microscopic features with macroscopic features.

DETAILED DESCRIPTION:
The overall objective of this study is to use VIO/FG-30350 ("VIO") to observe microscopic skin structure in people of different skin health at different anatomic locations and correlate microscopic features with macroscopic features.

ELIGIBILITY:
Inclusion Criteria:

Participants, ages 2 - 90 years old

Participant, or guardian, if applicable, must be willing to provide written informed consent prior to enrollment and agree to comply with protocol requirements. If applicable, child must be willing to provide written assent prior to enrollment and agree to comply with protocol requirements.

Participant or guardian, if applicable, must have sufficient mental capacity to understand the Informed Consent and provide clinically relevant and reliable feedback regarding their experience with the device.

Participant and guardian, if applicable, must comply with the protocol requirements.

Participant or guardian, if applicable, must agree that anonymized personal data will be made available to Study Sponsor and requisite regional and international regulatory bodies

Exclusion Criteria:

Any general health condition or systemic disease that may represent, in the opinion of the Principal Investigator, a potential increased risk associated with device use

Currently infected with a communicable skin infection (e.g., shingles or methicillin-resistant S. aureus), which does not include local and minimally pathogenic or non-pathogenic infections distant from the imaging location(s) (e.g., warts, acne)

Any known allergies to any materials used in the preparation of skin and/or device use

Has a temporary or permanent electrical implanted medical device

-

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Recruitment Clinics and Healthy Participants
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Correlational relationship | 7 days
  Correlational relationship of:
  melanin content quantified from noninvasive VIO images with
  macroscopic skin tone as measured with a colorimeter.
Correlational relationship | 7 days
  Correlational relationship of:
  1. melanin content quantified from noninvasive VIO images with
  2. macroscopic skin tone as measured with a colorimeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Enspectra Health, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: No